CLINICAL TRIAL: NCT05955105
Title: A Phase Ib/IIa, Multicenter, Open-label Study of ILB2109 and Toripalimab in Patients With Advanced Solid Malignancies
Brief Title: A Study of ILB2109 and Toripalimab in Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innolake Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILB2109A102
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer; Cervical Cancer; Endometrial Cancer; Triple Negative Breast Cancer; Ovarian Cancer; Soft Tissue Sarcoma; Melanoma; Nasopharyngeal Carcinoma; Non Small Cell Lung Cancer; Classic Hodgkin Lymphoma
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Sarcoma; Melanoma; Nasopharyngeal Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive ILB-2109 tablets and Toripalimab injection
  Interventions: Drug: ILB-2109; Drug: Toripalimab

INTERVENTIONS:
Drug: ILB-2109 — ILB-2109 tablets will be administered by mouth every day in 21-day cycles
Drug: Toripalimab — Toripalimab injection will be administered via IV every 21 days.

SUMMARY:
This is a multicenter, open-label, phase Ib/IIa study. The first part of the study will evaluate the safety, tolerability and preliminary efficacy of ILB2109 and Toripalimab in patients with locally advanced or metastatic solid malignancies. The second part of the study will evaluate the efficacy of ILB2109 and Toripalimab in patients with selected advanced solid malignancies.

DETAILED DESCRIPTION:
This is a two-part study consists of dose escalation and expansion in selected indications. The dose escalation part adopts a 3+3 protocol design and consists of 2 cohorts. Based on the data obtained from the escalation study, selected dose cohort will be expanded in 10 tumor types to further investigate the efficacy of the combination therapy. Subjects will be assessed for safety and efficacy outcomes at pre-specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between the ages of 18 and 80 years.
2. Patients with histologically or cytologically confirmed solid tumours that are advanced, metastatic and or progressive, for whom there is no effective standard therapy available.
3. Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤2.
4. Expected life expectancy ≥3 months.
5. Evaluable disease, either measurable on imaging, or with informative tumour marker(s), as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Eisenhauer, et al. 2009).
6. Laboratory values at Screening:

   Absolute neutrophil count ≥1.5 x 109/L; Platelets ≥75 x 109/L; Hemoglobin ≥ 90g/L; Total bilirubin <1.5 times the upper limit of normal; Aspartate aminotransferase (AST) ≤3 times the upper limit of normal, ≤ 5 times the upper limit of normal if subject has hepatic malignancies; Alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal, ≤ 5 times the upper limit of normal if subject has hepatic malignancies; Estimated glomerular filtration rate (GFR) of >50 mL/min (based on the Cockcroft-Gault formula; International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) ≤1.5 times the upper limit of normal; Left Ventricular Ejection Fraction (LVEF) ≥ 50%; Corrected QT Interval by Fridericia Method: male<450ms, female<470ms; and
7. Negative human chorionic gonadotropin (hCG) test in women of childbearing potential.
8. Sexually active male and female patients of childbearing potential must agree to use an effective method of birth control (e.g. barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices) during the entire duration of the study and for 90 days after final administration of ILB-2109, or the patient must be surgically sterile .
9. Ability to give written, informed consent prior to any study-specific Screening procedures.

Exclusion Criteria:

1. In the past 3 weeks: received systemic anti-tumor therapy, including chemotherapy, radiation, biologics, androgen, targeted therapy and immunotherapy with the following exceptions: i. received treatment containing nitrosoureas or mitomycin C in the past 6 weeks; ii. received oral fluorouracil or small molecule targeted therapy or Chinese Traditional Medicine (CTM) with anti-neoplasm indication in the past 2 weeks ;
2. In the past 4 weeks: received any other investigational treatment;
3. Gastrointestinal disease (e.g. Crohn's disease, ulcerative colitis, or short gut syndrome) that would impact on drug absorption;
4. Uncontrollable third-spacing of fluids;
5. Known CNS metastasis with clinical symptoms or the need of steroid treatment or CNS lesion ≥ 1.5cm or with the evidence of lesion enlargement in the past 4 weeks;
6. Severe cardiovascular diseases including symptomatic heart failure (NYHA Class II and above), unstable angina, arrythmia, myocardial infarction within the past 6 months, embolism or pulmonary embolism within the past 3 months;
7. Having any risk factors of QT prolongation, including present or family history of long QT syndrome or using any medication with known QT prolongation effect;
8. Poor controlled chronic diseases, including poorly controlled diabetes mellitus (defined as HbA1c ≥ 8.5%), poorly controlled hypertension, has a history of hypertensive emergency or hypertensive encephalopathy, endocrine diseases that require systemic therapy;
9. Current diagnosis of interstitial pneumonia or a history of chronic emphysema, COPD, or TB infection;
10. Autoimmune diseases that required systemic therapy within the past 2 years, with the exception of vitiligo, asthma, atopic diseases and autoimmune thyroid diseases that are stable on thyroid replacement therapy;
11. Active infection with the need if IV antibiotic treatment;
12. Known HIV infection;
13. Active HBV infection (defined as positive HBsAg and HBV-DNA>500 IU/ml), active HCV infection (positive HCV antibody but HCV-RNA < lower limit of detection is allowed to participate);
14. Known syphilis infection;
15. Received systemic steroid at a dose greater or equivalent to 10mg of prednisone per day or other immune modulating treatments in the past 14 days;
16. Plan to receive live vaccine during the study period (4 weeks prior to the 1st dose till 6 months after the last dose);
17. Major surgery within the past 4 weeks;
18. Previous allogeneic bone marrow transplant or solid organ transplant;
19. Known history of psychiatric disease/alcohol or drug abuse that would affect subject's compliance to trial protocol;
20. Any unresolved toxicities from prior therapies higher than CTCAE grade 1 with the following exceptions: i. alopecia; ii. peripheral neuropathy; iii. thyroid function abnormalities that can be treated with replacement therapy;
21. Known history of CTCAE grade 3 and above irAE in previous immunotherapies;
22. Known allergy to ILB-2109 or Toripalimab;
23. Subjects who are currently pregnant or breastfeeding;
24. Other conditions that in the opinion of the investigator will make the subject unfit to participate in this trial;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
The Incidence of DLTs | Cycle 1 (21 days)
  The incidence rate of Dose Limiting Toxicities (DLTs)
MTD | 6 months
  Determine the maximum tolerated dose (MTD) of ILB-2109 tablets
RP2D | 6 months
  Determine the recommended phase 2 dose (RP2D) when used in combination with Toripalimab for subsequent studies
The Objective Response Rate (ORR) | 36 months
  Observe the Objective Response Rate (ORR) of ILB-2109 tablets combined with Toripalimab in prespecified cohorts

SECONDARY OUTCOMES:
AE/TEAE/drug-related TEAE/irAE/SAE | 36 months
  Incidence of AE/TEAE/drug-related TEAE/irAE/SAE graded by CTCAE 5.0
Lab Abnormalities | 36 months
  Incidence of lab/physcial/EKG/vitals abnormalities graded by CTCAE 5.0
Peak Plasma Concentration (Cmax) | 36 months
  Study the Peak Plasma Concentration of ILB-2109 tablets
Area under the plasma concentration versus time curve (AUC) | 36 months
  Study the Area under the plasma concentration versus time curve (AUC) of ILB-2109 tablets
Half Life (T1/2) | 36 months
  Study the Half Life (T1/2) of ILB-2109 tablets
Time to maximum plasma concentration (Tmax) | 36 months
  Study the Time to maximum plasma concentration (Tmax) of ILB-2109 tablets
Clearance (CL) | 36 months
  Study the Clearance (CL) of ILB-2109 tablets
Volume of Distribution (Vd) | 36 months
  Study the Volume of Distribution (Vd) of ILB-2109 tablets
Progression Free Survival (PFS) | 36 months
  Observe the Progression Free Survival (PFS) in prespecified cohorts
Overall Survival (OS) | 36 months
  Observe the Overall Survival (OS) in prespecified cohorts
Duration of Response (DOR) | 36 months
  Observe the Duration of Response (DOR) in prespecified cohorts
Disease Control Rate (DCR) | 36 months
  Observe the Disease Control Rate (DCR) in prespecified cohorts
Time to Progression (TTP) | 36 months
  Observe the Time to Progression (TTP) in prespecified cohorts

OTHER OUTCOMES:
pCREB level in PBMC | 36 months
  Study the pharmacodynamic characteristics of ILB-2109 tablets, including the relationship between drug plasma concentration and the level of pCREB in PBMC.
Expression level of Adnosine Signature gene panel | 36 months
  Investigate potential biomarkers including the expression level of AdenoSig in tumor tissues
Tumor Mutational Burden | 36 months
  Investigate potential biomarkers including the TMB in tumor tissues
MSI Status | 36 months
  Investigate potential biomarkers including the MSI status in relationship to efficacy outcomes
PD-L1 | 36 months
  Investigate potential biomarkers including the expression level of PD-L1 in tumor tissues
CD68 | 36 months
  Investigate potential biomarkers including the expression level of CD68 in tumor tissues
A2aR | 36 months
  Investigate potential biomarkers including the expression level of A2aR in tumor tissues
CD8 | 36 months
  Investigate potential biomarkers including the expression level of CD8 in tumor tissues

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China